CLINICAL TRIAL: NCT00999830
Title: Randomised Phase II Study Evaluating the Anti-tumour Activity, Safety and Pharmacology of Two Dose Regimens of IPH2101, a Human Monoclonal Anti-KIR Antibody, in Patients With Multiple Myeloma in Stable Partial Response After a First Line Therapy
Brief Title: Evaluation of Activity, Safety and Pharmacology of IPH2101 a Human Monoclonal Antibody in Patients With Multiple Myeloma
Acronym: REMYKIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPH2101-201; NCT01937741 (obsolete NCT alias)
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2014-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — IPH-2101

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IPH 2101 0.2 mg/kg (Experimental): One infusion of IPH2101 every 4 weeks at the dose of 0.2 mg/kg by intravenous route over 1 hour, for 4 or up to 8 cycles.
  Interventions: Drug: IPH2101
- IPH2101 2.0 mg/kg (Experimental): One infusion of IPH2101 every 4 weeks at the dose of 2 mg/kg by intravenous route over 1 hour, for 4 or up to 8 cycles.
  Interventions: Drug: IPH2101

INTERVENTIONS:
Drug: IPH2101 — One infusion of IPH2101 every 4 weeks
  Other Names: Fully human anti-KIR monoclonal antibody (1-7F9)

SUMMARY:
This is an open randomised phase II study evaluating the anti-tumour activity, safety and pharmacology of two dose regimens of IPH2101, a human monoclonal anti-KIR antibody, in patients with multiple myeloma in stable partial response after a first line therapy.

DETAILED DESCRIPTION:
Development of new treatments for diseases such as multiple myeloma is a focus for research. The research being conducted is on treatment called Anti-KIR, which activates the body's own cells to kill tumor cells. This is different from many other treatments where chemicals are given to kill tumor cells.The primary objective of the study is to evaluate the clinical activity of two different dose regimens (0.2 mg/kg, leading to an intermittent saturation of NK receptors and 2mg/kg leading to a sustained saturation of NK receptors) of IPH2101 administered as a single agent in multiple myeloma patients who achieved, after the completion of any first line treatment, including conventional or high dose chemotherapies, a stable partial or very good partial response (PR or VGPR).

ELIGIBILITY:
Inclusion Criteria:

1. MM which initially required a systemic therapy and received a first line treatment, conventional doses of chemotherapies or high dose chemotherapy and an autologous transplantation of hematopoietic cells, followed or not by a consolidation treatment.
2. Residual disease considered as evaluable with:

   * Quantifiable serum M-protein: ≥ 3 g/l, except for spike in the beta globulin area. In this particular case serum M-protein is considered quantifiable if ≥ 10g/l
   * If serum M-protein is < 3g/l, measurable involved Free Light Chains ≥ 100 mg/l and an abnormal Free Light chains ratio (<0.26 or > 1.65)
3. Responses which are partial (PR and VGPR) and in plateau

   * Partial response should meet the IMWG uniform response criteria: a ≥ 50% reduction from value of serum M-protein before the first line chemotherapy treatment and a reduction in 24h urinary M-protein by ≥ 90% or to < 200 mg /24h;
   * Very good partial response according to the IMWG uniform response criteria with 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg/24h; furthermore the M-protein should spike in the gamma globulin area;
   * Plateau phase is defined by :

     * For patients with serum M-protein ≥ 3g/l: stable levels of M-protein in serum during at least 2 months checked on at least 3 consecutive samples, with the third evaluation performed within 4 weeks before study entry. Fluctuations of ± 25 % and ± 2 g/l in Serum M-protein levels are allowed.
     * For Patients with serum M-protein < 3g/l: stable levels Free Light Chains in serum during at least 2 months checked on at least 3 consecutive samples, with the third evaluation performed within 4 weeks before study entry. Fluctuations of ± 25 % of involved serum Free Light Chain are allowed.
4. ECOG performance status of 0, 1 or 2.
5. Clinical laboratory values at screening:

   * Calculated creatinine clearance (according to MDRD) > 50 ml/min
   * Platelet > 50 x 109 /l
   * ANC > 1 x 109 /l
   * Bilirubin levels < 1.5 ULN; ALT and AST < 2.5 ULN
6. Male or female patient who accepts and is able to use recognised effective contraception (oral contraceptives, IUCD, barrier method of contraception in conjunction with spermicidal jelly) throughout the study.
7. Signed inform consent obtained before any trial-related activities

Exclusion Criteria:

1. Age < 18 years old or > 75 years old
2. Previous consolidation/ maintenance therapy by Imid (thalidomide, lenalidomid) or bortezomib within the last 2 months
3. Treatment with chemotherapy, systemic corticosteroid within the previous 2 months
4. Treatment with growth factors (EPO, G- or GM-CSF) within the previous 1 month
5. Radiotherapy for bone or visceral lesion within the last 3 months
6. Use of any investigational agent within the last 2 months
7. Primary or associated amyloidosis
8. Peripheral neuropathy of grade ≥ III according to the CTCAE of the NCI
9. Abnormal cardiac status with any of the following

   1. NYHA stage III or IV congestive heart failure
   2. myocardial infarction within the previous 6 months
   3. symptomatic cardiac arrhythmia despite treatment
10. Current active infectious disease or positive serology for HIV, HCV or positive Hbs Antigen
11. History of or current auto-immune disease
12. Serious concurrent uncontrolled medical disorder
13. History of other malignancy for less then 5 years (apart from basal cell carcinoma of the skin, or in situ cervix carcinoma)
14. History of allogenic hematopoietic cell or solid organ transplantation
15. Pregnant or lactating women
16. Any medical condition which is regarded by the investigator as incompatible with the study participation
17. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel ATTAL, MD, Principal Investigator — University Hospital, Toulouse
Locations (9):
- France (9):
  - C.H.R.U. de Caen - Hôpital Bretonneau, Caen
  - CHU Dijon, Dijon
  - CHRU Lille, Lille
  - Hôpital Dupuytren, Limoges
  - Institut Paoli Calmettes, Marseille
  - CHU Nancy, Nancy
  - Hopital Saint Louis, Paris
  - Hôpital Saint Antoine, Paris
  - C.H.R.U. de Tours, Tours

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in France at the public hospital (10 actives center), from mid of November 2009 to end of October 2011.
Pre-assignment Details: All patients enrolled in the study were analyzed. There was no screen failure during the trial conduct.
Groups:
- Arm A: IPH2101 0.2mg/Kg: IPH2101 Fully human anti-KIR monoclonal antibody : 0.2mg/Kg , every 4 weeks by intravenous route over 1 hour, for 4 cycles. Patients responding at 4 months will be allowed to receive an additional period of treatment of 4 monthly.
- Arm B: IPH2101 2mg/kg: IPH2101 Fully human anti-KIR monoclonal antibody : 2mg/Kg , every 4 weeks by intravenous route over 1 hour, for 4 cycles. Patients responding at 4 months will be allowed to receive an additional period of treatment of 4 monthly.
Period: Overall Study
Arm/Group | Arm A: IPH2101 0.2mg/Kg | Arm B: IPH2101 2mg/kg
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: IPH2101 0.2mg/Kg; Arm B: IPH2101 2mg/kg: every 4 weeks by intravenous route over 1 hour, for 4 or up to 8 cycles.
- Total: Total of all reporting groups
Arm/Group | Arm A: IPH2101 0.2mg/Kg | Arm B: IPH2101 2mg/kg | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (5.6) | 55.9 (10.2) | 57.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 11 | 7 | 18
Region of Enrollment [Number; unit: participants]
  France | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Rate of Patients Achieving a Response Based on M-protein or Free Light Chains
Description: Response was defined:
  * In patients with a serum M-protein > 5 g/l, as a reduction of at least 25% (minor response according to European society for Blood and Marrow Transplantation (EBMT)) from baseline of serum M-protein confirmed on two consecutive determinations at 4 weeks interval;
  * In patients with a serum M-protein ≤ 5 g/l and ≥ 3g/l, as a negative electrophoresis
  * In patients with serum M-protein < 3 g/l but a measurable involved serum free light chains ≥ 100 mg/l and an abnormal Free Light Chains ratio (<0.26 or > 1.65), as a ≥ 50 % decrease in the difference between involved and uninvolved Free Light Chains levels.
Time Frame: From the start of the treatment to the End of Study and during the post study follow up during 2 years according to standard practices
Measure: Number; unit: participants
Arm/Group | Arm A: IPH2101 0.2mg/Kg | Arm B: IPH2101 2mg/kg
Number analyzed (Participants) | 14 | 13
participants | 0 | 1

2. Secondary Outcome: Biological Activity of IPH2101 on Killer Immunogloblin Like Receptors (KIR) Occupancy at End of Treatment
Description: KIR-occupancy is a relative measure of the fraction of cell surface KIR that is occupied by the IPH2101 monoclonal antibody, and hence is unavailable for binding to HLA ligands.
Time Frame: From the start up to the end of study (15 months)
Measure: Median (Full Range); unit: % of occupancy
Arm/Group | Arm A: IPH2101 0.2mg/Kg | Arm B: IPH2101 2mg/kg
Number analyzed (Participants) | 14 | 13
% of occupancy | 80.5 [33.8 to 95] | 96.8 [93 to 99.4]

3. Secondary Outcome: Safety Assessment
Description: Adverse Events, Serious Adverse Events, physical examination and biological changes.
Time Frame: from screening visit to the End of Study (at each study visit)
Measure: Number; unit: participants
Arm/Group | Arm A: IPH2101 0.2mg/Kg | Arm B: IPH2101 2mg/kg
Number analyzed (Participants) | 14 | 13
participants | 14 | 11

ADVERSE EVENTS:
Time Frame: Adverse events collected from screening visit (date of signature of Inform Consent Form) up to the End of Study
Arm/Group | Arm A: IPH2101 0.2mg/Kg | Arm B: IPH2101 2mg/kg
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/13
Other Adverse Events (participants affected / at risk) | 14/14 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: IPH2101 0.2mg/Kg (N=14) | Arm B: IPH2101 2mg/kg (N=13)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — This serious adverse event was not related to the investigational Medicinal Product
Disease progression (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: IPH2101 0.2mg/Kg (N=14) | Arm B: IPH2101 2mg/kg (N=13)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 4 (4) | 2 (2)
Fatigue (General disorders) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Chills (General disorders) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No